CLINICAL TRIAL: NCT00447408
Title: Impact of a PDA-Based Dietary Adherence Intervention on Interdialytic Weight Gain and Blood Pressure in Hemodialysis Patients
Brief Title: Impact of a Personal Digital Assistant (PDA) - Based Dietary Adherence Intervention on Interdialytic Weight Gain and Blood Pressure in Hemodialysis Patients
Acronym: BalanceWise-HD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Paul Teschan Research Fund (Other)
Responsible Party: Mary Ann Sevick, ScD, School of Medicine, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 0605006
Record Dates: First submitted 2007-03-12; First posted 2007-03-14 (Estimated); Last update posted 2010-06-28 (Estimated); Status verified 2010-06

CONDITIONS: End-Stage Renal Disease
Keywords: hemodialysis; dietary adherence; sodium
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Education in the hemodialysis diet.
  Interventions: Behavioral: Standard hemodialysis dietary instruction
- B (Experimental): Education in the hemodialysis diet. Behavioral counseling paired with PDA-based self-monitoring of dietary sodium intake.
  Interventions: Behavioral: Behavioral counseling plus PDA-based self-monitoring of diet

INTERVENTIONS:
Behavioral: Standard hemodialysis dietary instruction — Participants receive standard hemodialysis dietary instruction via a PowerPoint presentation delivered during routinely scheduled dialysis treatments.
  Arms: A
Behavioral: Behavioral counseling plus PDA-based self-monitoring of diet — Participants receive standard hemodialysis dietary instruction via a PowerPoint presentation delivered during routinely scheduled dialysis treatments. In addition they receive behavioral counseling paired with PDA-based self-monitoring of dietary sodium intake.
  Arms: B

SUMMARY:
With this study the investigators will test, in a randomised clinical trial (RCT), the efficacy of a behavioral dietary adherence enhancement intervention paired with PDA-based dietary self-monitoring for controlling sodium intake. Seventy hemodialysis patients will be recruited from units in Pittsburgh, Pennsylvania. Participants will be randomized to a 4-month PDA-based dietary counseling intervention or to a 4-month attention control. Potential participants will be stratified by whether or not they have diabetes. Data on primary and secondary outcomes will be obtained at baseline and four months. Primary dependent variables are:

1. adherence to dietary sodium targets as assessed from 3-day food recalls,
2. average monthly interdialytic weight gain, and
3. average pulse pressure. Secondary dependent variables are:
4. adherence to dietary targets for calories, protein, carbohydrates, fats, saturated fats, potassium, and phosphorus, as assessed from 3-day food recalls, (5) serum potassium and phosphorus levels determined on a monthly basis, and (6) nutritional status as determined from serum albumin. Laboratory data, interdialytic weight gain, and blood pressure data will be obtained per dialysis center routine and abstracted from the medical record. Three-day food recalls will be obtained at baseline, 4 and 8 months and analyzed using the Nutrient Data System.

ELIGIBILITY:
Inclusion Criteria:

* Those individuals who are 21 years of age or older
* Literate
* Community-dwelling adults
* Receiving maintenance HD for at least 3 months

Exclusion Criteria:

* Individuals who cannot read or write
* Those who do not speak English
* Those who plan to move out of the area or change dialysis centers within the next 6 months
* Those with a terminal illness and life expectancy of less than 12 months
* Those who are scheduled for a living donor transplant
* Individuals who cannot see the PDA screen or use the stylus to make selections from the PDA screen.
* Those individuals with a score ≤ 26 on the Mini Mental Status Exam.
* Also excluded will be individuals who are living in a nursing home or personal care facility, who would have limited control over their dietary intake.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2007-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
adherence to dietary sodium targets as assessed from 3-day food recalls | baseline and 4 months
average daily interdialytic weight gain (IDWG) | IDWG gathered with each dialysis treatment
average pulse pressure from pre-dialysis blood pressures | with each dialysis treatment

SECONDARY OUTCOMES:
adherence to dietary targets for calories, protein, carbohydrates, fats, saturated fats, potassium, and phosphorus, as assessed from 3-day food recalls | collected at baseline and 4 months
serum potassium and phosphorus levels | baseline, and 1, 2, 3, and 4 months
nutritional status as determined from serum albumin | baseline, 1, 2, 3, and 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Mary A Sevick, ScD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Campbell ZC, Dawson JK, Kirkendall SM, McCaffery KJ, Jansen J, Campbell KL, Lee VW, Webster AC. Interventions for improving health literacy in people with chronic kidney disease. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD012026. doi: 10.1002/14651858.CD012026.pub2. PMID 36472416